CLINICAL TRIAL: NCT06413693
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND (SPONSOR-OPEN) PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFECT OF PF-07293893 ON SKELETAL MUSCLE BIOMARKERS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A STUDY TO LEARN HOW THE STUDY MEDICINE CALLED PF-07293893 AFFECTS MUSCLE BIOMARKERS OF HEALTHY ADULTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5171004
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Healthy adult participants will receive a single dose of PF-07293893 or placebo
  Interventions: Drug: PF-07293893; Drug: Placebo
- Optional Cohort 2 (Experimental): Healthy adult participants will receive a single dose of PF-07293893 or placebo
  Interventions: Drug: PF-07293893; Drug: Placebo

INTERVENTIONS:
Drug: PF-07293893 — A single dose of PF-07293893 administered orally as tablets
Drug: Placebo — A single dose of Placebo administered orally as tablets that look the same as PF-07293893

SUMMARY:
The purpose of this study is to understand how the study medicine (PF-07293893) affects muscle biomarkers. Biomarkers are like clues or signs in our body that can help doctors understand our health. PF-07293893 is being studied as a possible treatment for people with heart disease who have reduced ability to exercise. This study aims to see how the study medicine affects muscle biomarkers related to the ability to exercise.

This study is seeking participants who:

1. Are males 18 to 65 years of age and females who are not able to become pregnant;
2. Have body mass index of 16 to 32 kilograms per meter square and a total body weight of more than 50 kilograms (110 pounds);
3. Over prior 4 weeks have an average of less than:

   -150 minutes of moderate-intensity aerobic physical activity throughout each week. Moderate-intensity physical activity feels somewhat hard. Your breathing becomes faster, but you are not out of breath. You can hold a conversation, but you cannot sing.

   AND

   -75 minutes of vigorous-intensity aerobic physical activity throughout each week. Vigorous-intensity physical activity feels challenging. You are breathing fast and deep. You cannot say more than a few words without pausing.

   OR

   -An equivalent combination of moderate-and vigorous-intensity activity.

   Participants will stay at the study clinic for about four days. On the third day, participants will take the study medicine or placebo (dummy pill) by mouth once at the study clinic and then stay at the study clinic for another day. During this time, the study team will check the treatment and take some blood and muscle tissue samples from the leg. This will help to understand if the study medicine affects muscle biomarkers. Participants will return to the study clinic for a follow-up visit or receive a follow-up telephone call about a month later.

ELIGIBILITY:
Inclusion Criteria:

1. Males 18 to 65 years of age and females of non-childbearing potential;
2. Body mass index (BMI) of 16 to 32 kg/m2; and a total body weight >50 kg (110 lb);
3. Over prior 4 weeks an average of less than 150 minutes of moderate-intensity aerobic physical activity throughout each week, and less than 75 minutes of vigorous-intensity aerobic physical activity throughout each week, or an equivalent combination of moderate- and vigorous-intensity activity.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease;
2. History of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C;
3. Kidney impairment as defined by an estimated glomerular filtration rate (eGFR) <75 mL/min/1.73 m²;
4. A positive urine drug test;
5. Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of skeletal muscle pACC/tACC ratio | Day 1 Pre-dose and 2 & 4 hours Post-dose

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events (AEs) | Baseline through Day 36
Number of Participants with change from Baseline in Laboratory Test Results | Baseline through Day 36
Number of Participants with Clinically Significant Change From Baseline in Vital Signs | Baseline through Day 36
Number of Participants with Clinically Significant Change From Baseline in 12-lead Electrocardiograms (ECGs) | Baseline and Day 1 Pre-dose and 6 hours Post-dose
Number of Participants With Change From Baseline in Physical Examinations | Baseline through Day 36
Maximum Observed Plasma Concentration (Cmax) | Day 1 Pre-dose, 0.5, 1, 2, 4, 6, 8 & 12 hours Post-dose and Day 2
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1 Pre-dose, 0.5, 1, 2, 4, 6, 8 & 12 hours Post-dose and Day 2
Area under the serum concentration vs. time curve for 0-24 hours (AUC24) | Day 1 Pre-dose, 0.5, 1, 2, 4, 6, 8 & 12 hours Post-dose and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Research Centers of America, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5171004